CLINICAL TRIAL: NCT02016079
Title: Randomized Controlled Trial of Omega-3 on Child Behavior Problems
Brief Title: Effect of Omega-3 Supplementation on Child Behavior Problems
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joint Child Health Project, Mauritius (Other)
Responsible Party: Principal Investigator, Tashneem Moohamed, National Director, JCHP, Joint Child Health Project, Mauritius
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JCHP-01; JCHP-N3 (Other: JCHP)
Record Dates: First submitted 2013-12-10; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Antisocial; Aggressive; Externalizing Behavior Problems; Internalizing Behavior Problems
Keywords: randomized controlled trial; omega-3; nutrition; behavior problems; externalizing; internalizing; antisocial; aggressive
MeSH Terms: conditions — Antisocial Personality Disorder; Aggression; Mental Disorders | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 (Experimental): a fruit drink containing omega-3
  Interventions: Dietary Supplement: omega-3
- Fruit drink (Placebo Comparator): the same fruit drink given in the experimental arm, but not containing omega-3

INTERVENTIONS:
Dietary Supplement: omega-3 — 200 ml fruit drink containing omega-3
  Other Names: Smartfish
  Arms: Omega-3

SUMMARY:
The primary purpose of this study was to assess the effectiveness of omega-3 supplementation on behavior problems in children.

DETAILED DESCRIPTION:
This study consists of a randomized, placebo-controlled, double-blind trial of omega-3 on behavior problems in children. All behavior problem outcomes were assessed, although the primary focus was on antisocial and aggressive behavior.

ELIGIBILITY:
Inclusion Criteria:

* child
* age between 8 and 16 years
* residing in the community

Exclusion Criteria:

* fish allergy
* diagnosed mental disorder
* mental retardation
* on medication that may modify lipid metabolism
* extensive use of nutritional supplements within the previous 3 months

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist | 6 months
  The outcome measure assessed internalizing and externalizing behavior problems in children
Reactive-Proactive Aggression Questionnaire | 6 months
  A self-report measure of reactive and proactive forms of aggressive behavior
Antisocial Personality Screening Device | 6 months
  A measure of antisocial personality, with a total score and three subscales: callous-unemotional, impulsivity, narcissism

SECONDARY OUTCOMES:
WISC | 6 months
  estimate of IQ

CONTACTS AND LOCATIONS:
Overall Officials: Tashneem Moohamed, BSc, Principal Investigator — Joint Child Health Project; Cyril Dalais, MSc, Principal Investigator — Action Research Program, Educational Priroity Areas, Mauritius
Locations (1):
- Joint Child Health Project, Quatre Bornes, Mauritius

REFERENCES:
- [Derived] Raine A, Portnoy J, Liu J, Mahoomed T, Hibbeln JR. Reduction in behavior problems with omega-3 supplementation in children aged 8-16 years: a randomized, double-blind, placebo-controlled, stratified, parallel-group trial. J Child Psychol Psychiatry. 2015 May;56(5):509-20. doi: 10.1111/jcpp.12314. Epub 2014 Aug 22. PMID 25146492